CLINICAL TRIAL: NCT00482014
Title: Phase 1/2 Study of Pemetrexed (Alimta) Plus Carboplatin, or Pemetrexed Plus Cisplatin With Concurrent Radiation Therapy Followed by Every-21-Day Pemetrexed Consolidation in Patients With Favorable-Prognosis Inoperable Stage IIIA/B Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: A Study of Pemetrexed Plus Carboplatin, or Pemetrexed Plus Cisplatin With Radiation Therapy Followed by Pemetrexed in Patients With Inoperable Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9031; H3E-US-S047 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-10

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Pemetrexed + Carboplatin (Experimental): Pemetrexed + Carboplatin
  Interventions: Drug: pemetrexed; Drug: carboplatin; Radiation: radiation therapy
- B: Pemetrexed + Cisplatin (Experimental): Pemetrexed + Cisplatin
  Interventions: Drug: pemetrexed; Drug: cisplatin; Radiation: radiation therapy

INTERVENTIONS:
Drug: pemetrexed — Phase 1 - 500 milligram/meter squared (mg/m²), administered intravenously, every 21 days for 3 cycles
  Phase 2 - 500 mg/m², administered intravenously, every 21 days for 3 cycles
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation therapy for each phase
  Other Names: LY231514; Alimta
Drug: cisplatin — Phase 1 - 30 mg/m² and 75 mg/m², administered intravenously, Days 1, 8, 22, 29 and 43
  Phase 2 - 75 mg/m², administered intravenously, every 21 days for 3 cycles
  Arms: B: Pemetrexed + Cisplatin
Drug: carboplatin — Phase 1 - dosed at area under the curve (AUC) 2 milligram/milliliter*minute (mg/mL*min), administered intravenously, Days 1, 8, 22, 29 and 43
  Phase 2 - dosed at AUC 5 mg/mL*min, administered intravenously, every 21 days for 3 cycles
  Arms: A: Pemetrexed + Carboplatin
Radiation: radiation therapy — Phase 1 - 2 Gray, daily, 5 days a week for Days 1-51
  Phase 2 - 2 Gray, daily, 5 days a week for Days 1-45

SUMMARY:
The primary purpose of this study is to determine the 2-year survival rate of both of the chemotherapy regimens in patients with inoperable non-small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable non small cell lung cancer
* No weight loss greater than 10% in 3 months prior to enrolling in trial
* Adequate kidney function
* Adequate liver function
* Adequate lung function

Exclusion Criteria:

* Previous surgery to remove lung tumor
* Previous chemotherapy or radiation therapy or lung cancer
* Inability to take vitamin supplementation
* Heart attack within past 6 months
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corpus Christi, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Temple, Texas
- India (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Carboplatin (Study Phase 1): 500 milligrams/meter squared (mg/m²) pemetrexed (Pem) every 21 days for 3 cycles + Carboplatin (Carbo) dosed at area under the curve (AUC) 2 milligram/milliliter*minute (mg/mL*min) on Days 1, 8, 22, 29, 43 + radiation therapy (RT) 74 Grays (Gy) total dose given 2 Gy/day over 51 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Carbo + RT) therapy.
- Pemetrexed + Cisplatin (Study Phase 1): 500 mg/m² pemetrexed every 21 days for 3 cycles + Cisplatin (Cis) 30 mg/m² or 75 mg/m² on Days 1, 8, 22, 29, 43 + radiation therapy 74 Gy total dose given 2 Gy/day over 51 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Cis + RT) therapy.
- Pemetrexed + Carboplatin (Study Phase 2): 500 mg/m² pemetrexed every 21 days for 3 cycles + Carboplatin dosed at AUC 5 mg/mL*min every 21 days for 3 cycles + radiation therapy 64-68 Gy total dose given 2 Gy/day over 45 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Carbo + RT) therapy.
- Pemetrexed + Cisplatin (Study Phase 2): 500 mg/m² pemetrexed every 21 days for 3 cycles + Cisplatin 75 mg/m² every 21 days for 3 cycles + radiation therapy 64-68 Gy total dose given 2 Gy/day over 45 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Cis + RT) therapy.
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin (Study Phase 1) | Pemetrexed + Cisplatin (Study Phase 1) | Pemetrexed + Carboplatin (Study Phase 2) | Pemetrexed + Cisplatin (Study Phase 2)
Started | 9 | 13 | 46 | 52
Completed | 2 | 7 | 35 | 29
Not Completed | 7 | 6 | 11 | 23
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 4
Not completed — Adverse Event | 3 | 0 | 2 | 8
Not completed — Death | 1 | 2 | 1 | 4
Not completed — Lack of Efficacy | 1 | 0 | 4 | 6
Not completed — Sponsor Decision | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Carboplatin (Study Phase 1) | Pemetrexed + Cisplatin (Study Phase 1) | Pemetrexed + Carboplatin (Study Phase 2) | Pemetrexed + Cisplatin (Study Phase 2) | Total
Number analyzed (Participants) | 9 | 13 | 46 | 52 | 120
Age Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (8.70) | 61.0 (11.66) | 63.6 (9.92) | 64.1 (9.44) | 63.4 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 16 | 21 | 43
  Male | 7 | 9 | 30 | 31 | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 8 (73.3) | 7 | 36 | 37 | 88
  African | 1 (11.7) | 3 | 5 | 5 | 14
  Hispanic | 0 (1.7) | 1 | 1 | 0 | 2
  East Asian | 0 (1.7) | 0 | 1 | 1 | 2
  West Asian (Indian sub continent | 0 (11.7) | 2 | 3 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 9 | 13 | 43 | 43 | 108
  India | 0 | 0 | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of Carboplatin
Description: MTD was defined as a dose at which the occurrence of at least 2 dose-limiting toxicities (DLTs) was observed. DLT was defined as any of the following events occurring during the entire radiation therapy (RT) course, including a 2-week recovery period following completion of RT: Grade 4 neutropenia (<0.5 x 10^9 cells per liter) lasting >7 days, febrile neutropenia; ≥Grade 3 neutropenia with fever >38.5 degrees Celsius (°C), Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with ≥Grade 2 bleeding, ≥Grade 3 nonhematologic toxicity (excluding nausea, vomiting, and transaminase elevations) and ≥Grade 3 pulmonary or esophageal toxicity (radiation-related pneumonitis or esophagitis).
Time Frame: Phase 1 enrollment to the end of study treatment up to Week 11
Population: All participants who were enrolled in Study Phase 1 and completed at least 6 weeks of pemetrexed + carboplatin treatment.
Measure: Number; unit: milligram/milliliter*minute (mg/mL*min)
Groups:
- Pemetrexed + Carboplatin Treatment Group: 500 milligrams/meter squared (mg/m²) pemetrexed (Pem) every 21 days for 3 cycles + Carboplatin (Carbo) dosed at area under the curve (AUC) 2 milligram/milliliter*minute (mg/mL*min) on Days 1, 8, 22, 29, 43 + radiation therapy (RT) 74 Grays (Gy) total dose given 2 Gy/day over 51 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Carbo + RT) therapy.
Arm/Group | Pemetrexed + Carboplatin Treatment Group
Number analyzed (Participants) | 9
milligram/milliliter*minute (mg/mL*min) | NA — MTD was not reached because 2 DLTs threshold wasn't reached.

2. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of Cisplatin
Description: as for outcome 1
Time Frame: Phase 1 enrollment to the end of study treatment up to Week 11
Population: All participants who were enrolled in Study Phase 1 and completed at least 6 weeks of pemetrexed + cisplatin treatment.
Measure: Number; unit: milligrams/meter squared (mg/m²)
Groups:
- Pemetrexed + Cisplatin Treatment Group: 500 milligrams/meter squared (mg/m²) pemetrexed every 21 days for 3 cycles + Cisplatin (Cis) 30 mg/m² or 75 mg/m² on Days 1, 8, 22, 29, 43 + radiation therapy 74 Gy total dose given 2 Gy/day over 51 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Cis + RT) therapy.
Arm/Group | Pemetrexed + Cisplatin Treatment Group
Number analyzed (Participants) | 13
milligrams/meter squared (mg/m²) | NA — MTD was not reached because 2 DLTs threshold wasn't reached.

3. Secondary Outcome: Phase 1 - Pharmacology Toxicity: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Phase 1 pharmacology toxicity was defined as the number of participants experiencing dose limiting toxicities (DLTs). DLT was defined as any of the following events occurring during the entire radiation therapy (RT) course: Grade 4 neutropenia (<0.5 x 10^9 cells per liter) >7 days, febrile neutropenia, ≥Grade 3 neutropenia with fever >38.5 degrees Celsius (°C), Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with ≥Grade 2 bleeding, ≥Grade 3 nonhematologic toxicity (excluding nausea, vomiting, and transaminase elevations), and ≥Grade 3 pulmonary or esophageal toxicity (radiation-related pneumonitis or esophagitis). Grade 5 events are the events leading to the death.
Time Frame: Phase 1 enrollment up to Week 11
Population: All participants who were enrolled in Study Phase 1 and received at least 1 dose of study drug and 1 dose of radiation therapy.
Measure: Number; unit: participants
Groups:
- Pemetrexed + Cisplatin Treatment: 500 mg/m² pemetrexed every 21 days for 3 cycles + Cisplatin (Cis) 30 mg/m² or 75 mg/m² on Days 1, 8, 22, 29, 43 + radiation therapy 74 Gy total dose given 2 Gy/day over 51 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Cis + RT) therapy.
Arm/Group | Pemetrexed + Carboplatin Treatment Group | Pemetrexed + Cisplatin Treatment
Number analyzed (Participants) | 9 | 11
participants
  Grade 5 Pneumocystis jiroveci pneumonia | 1 | 0
  Grade 5 Hemoptysis (pemetrexed+Cisplatin30 mg/m² ) | 0 | 1

4. Secondary Outcome: Phase 1 - Percentage of Participants With Complete Response or Partial Response (Response Rate)
Description: Response rate is the percentage of participants with complete response (CR) or partial response (PR), as assessed according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. Response rate is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: Phase 1 enrollment to the end of the study treatment up to Week 11
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin Treatment Group | Pemetrexed + Cisplatin Treatment
Number analyzed (Participants) | 9 | 11
percentage of participants
  Complete Response (CR) | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Partial Response (PR) | 11.1 [0.28 to 48.25] | 45.5 [16.75 to 76.62]

5. Secondary Outcome: Phase 2 - Pharmacology Toxicity: Number of Participants With Adverse Events
Description: Phase 2 pharmacology toxicity was defined as the number of participants who experienced serious adverse events or all other nonserious adverse events during the study. A summary of serious adverse events and other nonserious adverse events is located in the Reported Adverse Events section.
Time Frame: Phase 2 randomization to the end of the study treatment up to 30.0 months
Population: All randomized participants who received at least 1 dose of study drug or 1 dose of radiation therapy (RT) during Study Phase 2.
Measure: Number; unit: participants
Groups:
- Pemetrexed + Carboplatin Treatment Group: 500 milligrams/meter squared (mg/m²) pemetrexed (Pem) every 21 days for 3 cycles + Carboplatin (Carbo) dosed at area under the curve (AUC) 5 milligram/milliliter*minute (mg/mL*min) every 21 days for 3 cycles + radiation therapy (RT) 64-68 (Gray) Gy total dose given 2 Gy/day over 45 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Carbo + RT) therapy.
- Pemetrexed + Cisplatin Treatment Group: 500 mg/m² pemetrexed every 21 days for 3 cycles + Cisplatin (Cis) 75 mg/m² every 21 days for 3 cycles + radiation therapy 64-68 Gy total dose given 2 Gy/day over 45 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Cis + RT) therapy.
Arm/Group | Pemetrexed + Carboplatin Treatment Group | Pemetrexed + Cisplatin Treatment Group
Number analyzed (Participants) | 46 | 52
participants
  Serious Adverse Events | 21 [6.0 to 12.6] | 19 [8.3 to NA]
  Other Nonserious Adverse Events | 44 | 51

6. Secondary Outcome: Phase 2 - Time to Progression
Description: Time to disease progression was measured from randomization of Study Phase 2 to the first observation of disease progression according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Disease progression is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Phase 2 randomization to measured disease progression up to 24 months
Population: All randomized participants in Study Phase 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin Treatment Group | Pemetrexed + Cisplatin Treatment Group
Number analyzed (Participants) | 46 | 52
months | 8.8 [6.0 to 12.6] | 13.1 [8.3 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

7. Secondary Outcome: Phase 2 - Median Survival
Time Frame: Phase 2 randomization to death as the result of any cause up to 30.0 month
Population: All randomized participants in Study Phase 2.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pemetrexed + Carboplatin Treatment Group: 500 milligrams/meter squared (mg/m²) pemetrexed (Pem) every 21 days for 3 cycles + Carboplatin (Carbo) dosed at area under the curve (AUC) 5 milligram/milliliter*minute (mg/mL*min) every 21 days for 3 cycles + radiation therapy (RT) 64-68 Gray (Gy) total dose given 2 Gy/day over 45 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Carbo + RT) therapy.
Arm/Group | Pemetrexed + Carboplatin Treatment Group | Pemetrexed + Cisplatin Treatment Group
Number analyzed (Participants) | 46 | 52
months | 18.7 [12.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 27.0 [23.2 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

8. Secondary Outcome: Phase 2 - Percentage of Participants With Complete Response or Partial Response (Response Rate)
Description: as for outcome 4
Time Frame: Phase 2 randomization to the end of the treatment up to 30.0 months
Population: All randomization participants in Study Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin Treatment Group | Pemetrexed + Cisplatin Treatment Group
Number analyzed (Participants) | 46 | 52
percentage of participants
  Complete Response (CR) | 6.5 [1.4 to 17.9] | 3.8 [0.5 to 13.2]
  Partial Response (PR) | 45.7 [30.9 to 61.0] | 42.3 [28.7 to 56.8]

9. Primary Outcome: Phase 2 - Survival Probability at 2 Years
Time Frame: Phase 2 randomization up to 2 years
Population: All randomized participants in Study Phase 2.
Measure: Mean (95% Confidence Interval); unit: percentage survival
Arm/Group | Pemetrexed + Carboplatin Treatment Group | Pemetrexed + Cisplatin Treatment Group
Number analyzed (Participants) | 46 | 52
percentage survival | 45.4 [29.5 to 60.0] | 58.4 [42.6 to 71.3]

ADVERSE EVENTS:
Groups:
- Phase 1: Pemetrexed + Carboplatin: 500 milligrams/meter squared (mg/m²) pemetrexed (pem) every 21 days for 3 cycles + Carboplatin (Carbo) dosed at area under the curve (AUC) 2 milligram/milliliter*minute (mg/mL*min) on Days 1, 8, 22, 29, 43 + radiation therapy (RT) 74 Grays (Gy) total dose given 2 Gy/day over 51 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Carbo + RT) therapy.
- Phase 1: Pemetrexed + Cisplatin: 500 mg/m² pemetrexed every 21 days for 3 cycles + Cisplatin (Cis) 30 mg/m² or 75 mg/m² on Days 1, 8, 22, 29, 43 + radiation therapy 74 Grays (Gy) total dose given 2 Gy/day over 51 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Cis + RT) therapy.
- Phase 2: Pemetrexed + Carboplatin: 500 mg/m² pemetrexed every 21 days for 3 cycles + Carboplatin dosed at AUC 5 mg/mL*min every 21 days for 3 cycles + radiation therapy 64-68 Gy total dose given 2 Gy/day over 45 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Carbo + RT) therapy.
- Phase 2: Pemetrexed + Cisplatin: 500 mg/m² pemetrexed every 21 days for 3 cycles + Cisplatin 75 mg/m² every 21 days for 3 cycles + radiation therapy 64-68 Gy total dose given 2 Gy/day over 45 days.
  Consolidation Therapy - 500 mg/m² pemetrexed, administered intravenously, every 21 days for 3 cycles beginning 3 weeks after completion of chemoradiation (Pem + Cis + RT) therapy.
Arm/Group | Phase 1: Pemetrexed + Carboplatin | Phase 1: Pemetrexed + Cisplatin | Phase 2: Pemetrexed + Carboplatin | Phase 2: Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 6/9 | 5/13 | 21/46 | 19/52
Other Adverse Events (participants affected / at risk) | 9/9 | 10/13 | 44/46 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Pemetrexed + Carboplatin (N=9) | Phase 1: Pemetrexed + Cisplatin (N=13) | Phase 2: Pemetrexed + Carboplatin (N=46) | Phase 2: Pemetrexed + Cisplatin (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — One of the events resulted in a discontinuation due to death.
Oedema peripheral (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — The event in Pemetrexed + Cisplatin resulted in a discontinuation due to death.
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This event resulted in a discontinuation due to death.
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (8)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — This event resulted in a discontinuation due to death.
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — The event in Pemetrexed + Cisplatin treatment group resulted in a discontinuation due to death.
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — This event resulted in a discontinuation due to death.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (7)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Pemetrexed + Carboplatin (N=9) | Phase 1: Pemetrexed + Cisplatin (N=13) | Phase 2: Pemetrexed + Carboplatin (N=46) | Phase 2: Pemetrexed + Cisplatin (N=52)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 5 (6) | 14 (24) | 16 (23)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 5 (6) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (5) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 16 (27) | 12 (15)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 4 (8) | 5 (7)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (Cardiac disorders) | 0 (0) | 1 (2) | 4 (6) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (6) | 14 (17) | 15 (16)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (7) | 10 (10)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 7 (8) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 6 (8) | 5 (5) | 19 (20) | 18 (25)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (7) | 21 (24) | 28 (40)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 19 (23) | 21 (26)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (3) | 8 (13) | 17 (24)
Asthenia (General disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (8)
Breakthrough pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 7 (7) | 7 (11)
Chills (General disorders) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Fatigue (General disorders) | 6 (7) | 7 (8) | 26 (32) | 27 (36)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 4 (6) | 5 (5)
Hypoalbuminaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (6)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 5 (5) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Blood creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blood lactate dehydrogenase (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 8 (12) | 4 (7)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (6) | 3 (4)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 4 (9) | 3 (4)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 13 (13) | 9 (9)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 12 (12) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (2) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 10 (10) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 6 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 10 (16) | 8 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (7) | 8 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 5 (5) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 9 (10) | 4 (7)
Dysgeusia (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5) | 5 (6)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 5 (5) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 6 (6) | 6 (6)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 6 (7) | 6 (6)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 11 (11) | 9 (9)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 15 (15) | 14 (16)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 9 (10) | 12 (13)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (5)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days